CLINICAL TRIAL: NCT04130386
Title: Motivational Interviewing to Address Freshman Weight Gain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Auburn University (Other)
Responsible Party: Principal Investigator, Danielle D Wadsworth, Associate Professor, Auburn University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AuburnU-MI college freshman
Record Dates: First submitted 2019-10-01; First posted 2019-10-17 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Motivational Interviewing
MeSH Terms: interventions — Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: Assigned to either motivational interviewing or e-education.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivational Interviewing (Experimental): Participants assigned to this arm will complete three MI sessions over 10 weeks.
  Interventions: Behavioral: Motivational Interviewing
- E-education (Active Comparator): The e-education group receives three educational modules lasting approximately 10 minutes each over a period of 10 weeks.
  Interventions: Behavioral: e-education

INTERVENTIONS:
Behavioral: Motivational Interviewing — Participants receiving MI
  Arms: Motivational Interviewing
Behavioral: e-education — Participants receiving e-education
  Arms: E-education

SUMMARY:
The purpose of the study is to determine the effect of Motivational Interviewing and e-health education on body composition and psychological outcomes. After baseline testing, participants will be randomly assigned to a motivational interviewing or e-health education group for a 10-week intervention. Variables of interest include: body composition, physical activity, food consumption and self-determination theory constructs.

ELIGIBILITY:
Inclusion Criteria:

1. Classified as a college freshman and 18 years of age.
2. Low risk for medical complications from exercise (as determined by physical activity readiness questionnaire (PARQ+).
3. Neither currently engaging in exercise nor consistently exercising over the last three months (2 days per week or less).
4. Be considered overweight based on BMI (BMI at or above 25)
5. Not pregnant.

Exclusion Criteria:

* Those that do not meet inclusion criteria.

Ages: 18 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
changes in fat mass | 12 and 28 weeks
  changes in fat mass measured in KG by a iDXA scan
Changes in lean mass | 12 and 28 weeks
  changes in lean mass measured in KG by a iDXA scan
Physical Activity | 12 and 28 weeks
  Changes in minutes of moderate to vigorous physical activity measured by an accelerometer.
Changes in the number of servings of Fruit and Vegetables | 12 and 28 weeks
  Changes in fruit and vegetable consumption measured in servings per day
Changes in Autonomous motivation | 12 and 28 weeks
  Changes in Autonomous motivation will be assessed with the Exercise Regulation Questionnaire (BREQ-3). The score range for each subscale is 0-16. A higher score for each subscales represents higher levels of motivation for external, introjected, identified and integrated forms of motivation.

SECONDARY OUTCOMES:
Experience with MI | 12 weeks
  Participants experience with the MI intervention will be assessed with the Health care climate questionnaire. This scale measures perceived autonomous support. The score ranges from 15-105, with higher scores associated with higher levels of perceived autonomy support.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Kinesiology, Auburn, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available

REFERENCES:
- [Derived] Suire KB, Kavookjian J, Strunk K, Wadsworth DD. Motivational interviewing for weight management among college students during COVID-19: An exploratory randomized controlled trial. Obes Pillars. 2023 Dec 26;9:100097. doi: 10.1016/j.obpill.2023.100097. eCollection 2024 Mar. PMID 38268522